CLINICAL TRIAL: NCT03643666
Title: Intraperitoneal Dexamethasone vs Dexamethasone Plus Magnesium Sulphate for Pain Relief in Laparoscopic cholecystectomY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdElKhalik Mahmoud Shaban, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-9-2018
Record Dates: First submitted 2018-08-20; First posted 2018-08-23 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): this group will include 25 patients receiving intraperitoneal 40 ml of normal saline only at the end of laparoscopic cholecystectomy
  Interventions: Drug: Placebo (saline)
- dexamethasone group (Active Comparator): this group will include 25 patients receiving intraperitoneal 16 mg dexamethasone in 40 ml saline at the end of laparoscopic cholecystectomy
  Interventions: Drug: dexamethasone
- dexamethasone plus magnesium sulphate group (Active Comparator): this group will include 25 patients receiving intraperitoneal 16 mg dexamethasone plus 2 gm magnesium sulphate at the end of laparoscopic cholecystectomy
  Interventions: Drug: dexamethasone; Drug: magnesium sulphate

INTERVENTIONS:
Drug: dexamethasone — before closure of the laparoscopic entering sites the patients will receive instillation of 40 ml of normal saline containing 16mg dexamethasone
  Arms: dexamethasone group; dexamethasone plus magnesium sulphate group
Drug: magnesium sulphate — patients will receive instillation of 40 ml of normal saline containing 16mg dexamethasone plus magnesium sulphate 2 gm into the peritoneum at the end of the operation
  Arms: dexamethasone plus magnesium sulphate group
Drug: Placebo (saline) — before closure of the laparoscopic entering sites the patients received instillation of 40 ml normal saline into the peritoneum
  Arms: control group

SUMMARY:
Laparoscopic cholecystectomy has become a standard technique for gall bladder surgery. Benefits in comparison to conventional laparotomy are shorter lived effects on pulmonary function and less postoperative pain . However, patients often suffer from considerable pain during the first 24 postoperative hours. Pain can prolong hospital stay and lead to increased morbidity, which is particularly important now that many centers are performing this operation as a day-case procedure. Administration of intraperitoneal local anesthetic, either during or after surgery, is used by as a method of reducing postoperative pain. Although a number of studies have reported a significant reduction in postoperative pain after the use of intraperitoneal analgesia, others have reported no benefit. Several investigations have been conducted in order to find the cause of this pain. According to some of these investigations, the pain is attributed to peritoneal inflammation due to carbon dioxide pneumoperitoneum. Since steroids have been used for reducing inflammation, they may be considered as alternatives for relieving pain. Dexamethasone is a strong long acting glucocorticoid and it is widely used after surgery. it has been established that steroids are effective in relieving postoperative pain in laparoscopic cholecystectomy. Also, administration of magnesium sulphate has been shown to have a potential to prevent postoperative pain and to reduce intra operative anesthetic and analgesic requirements being an antagonist of N-methyl-D-aspartate (NMDA) receptors and its associated ion channels. Some studies showed reduction of pain scores if magnesium sulphate was injected intra-articular and intraperitoneal with no serious adverse effects. In this study the investigators will use intraperitoneal dexamethasone vs dexamethasone plus magnesium sulphate to study their analgesic efficacy after laparoscopic cholecystectomy as the investigators assume that the combination of both drugs will provide stronger analgesia than dexamethasone alone

ELIGIBILITY:
Inclusion Criteria:

1. Age group and gender: between 18 to 60 years both males and females
2. American Society of Anesthesiologists (ASA) physical status I-II

Exclusion Criteria:

1. Age < 18 years or > 60 years
2. ASA physical status III or IV
3. Patients with diabetes
4. Patient refusal to participate in the study
5. Chronic respiratory disease
6. Advanced renal or hepatic diseases
7. Use of opioids, tranquilizers or steroids
8. Confusion or psychiatric illness
9. Acute cholecystectomy
10. Patients with peritoneal drain after surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain: VAS | first 24 hours
  Postoperative pain scoring using standard Visual Analogue Scale (VAS) pain score of 0-10 (with 0 meaning no pain and 10 meaning the most intense pain ever experienced)

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | first 24 hours
  Postoperative nausea and vomiting using simplified simplified postoperative nausea and vomiting (PONV) impact scale which is measured through two questions as following:
  Q1. Has the patient vomited or had dry-retching? 0. No
  1. Once
  2. Twice
  3. Three or more times Q2. Has the patient experienced a feeling of nausea (an unsettled feeling in the stomach and slight urge to vomit)? If yes, has the feeling of nausea interfered with activities of daily life, such as being able to get out of bed, being able to move about freely in bed, being able to walk normally, or eating and drinking?
  0. Not at all
  1. Sometimes
  2. Often or most of the time
  3. All of the time. To calculate the PONV Impact Scale, the numerical responses to questions 1 and 2 will be added. Several vomits or dry-retching events occurring over a short time frame e.g 5 min, will be counted as one vomiting/dry-retching episode.
Heart rate | first 24 hours
arterial blood pressure measurement postoperative | first 24 hours
  systolic and diastolic blood pressure
doses of consumed postoperative analgesics | first 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini hospital, Cairo, Egypt